CLINICAL TRIAL: NCT00968851
Title: A Randomized Double-Blind Placebo-Controlled 12-Week Phase 2 Study of Two Different Doses of an Alpha-7 Nicotinic Acetylcholine Receptor Agonist(EVP-6124)or Placebo in Schizophrenia Subjects on Chronic Stable Atypical Anti-Psychotic Therapy
Brief Title: Safety and Cognitive Function Study of EVP-6124 in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FORUM Pharmaceuticals Inc (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVP-6124-009
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2012-03

CONDITIONS: Schizophrenia; Central Nervous System Diseases; Cognition
Keywords: Schizophrenia; Central nervous System Diseases; Cognition
MeSH Terms: conditions — Schizophrenia; Central Nervous System Diseases | interventions — 7-chloro-N-quinuclidin-3-yl-benzo(b)thiophene-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- EVP-6124 0.3 mg (Active Comparator): one 0.3 mg capsule every day for 84 days
  Interventions: Drug: EVP-6124
- EVP-6124 1.0 mg (Active Comparator): one 1.0 mg capsule every day for 84 days.
  Interventions: Drug: EVP-6124
- Placebo (Placebo Comparator): Placebo every day for 84 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EVP-6124 — Arms: 1
  Arms: EVP-6124 0.3 mg
Drug: Placebo — Arm: 3
  Arms: Placebo
Drug: EVP-6124 — Arms: 2
  Arms: EVP-6124 1.0 mg

SUMMARY:
This study is being conducted to determine the safety and effect on cognitive function of two different doses of an investigational medication, EVP-6124, in individuals with schizophrenia who are on chronic stable atypical anti-psychotic therapy. In addition, behavioral and psychotic symptoms will be evaluated.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, Phase 2 safety/efficacy study in which two dose levels of EVP-6124 will be evaluated. Eligible for enrollment will be patients who meet clinical criteria for schizophrenia and who are taking chronic atypical anti-psychotic medication at a stable dose. This study will therefore evaluate the effects of EVP-6124 when administered concomitantly with anti-psychotic medication.

Patients will be randomized to one of the following groups: 0.3 mg or 1.0 mg EVP-6124, or placebo. Seventy-five patients per group. Study drug will be supplied as capsules and will be orally administered once daily for a total of 84 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet clinical criteria for schizophrenia or schizo-affective disorder utilizing the structured clinical interview (SCI)
* Must be treated with a second generation anti-psychotic drug other than clozapine at a stable dose for at least 4 weeks and must have been on that drug and clinically stable for at least 8 weeks
* Must have no more than "moderate" severity rating for negative symptoms: BPRS item ≤4
* A minimal level of extrapyramidal symptoms (EPS); Simpson-Angus Scale total score ≤6
* A minimal level of depression; Calgary Depression Scale total score ≤10
* Must have a general health status acceptable for participation in a 12-week clinical trial
* Fluency (oral and written) in the language in which the standardized tests will be administered
* If a smoker, the ability to refrain from smoking for at least 30 minutes prior to any cognitive testing

Exclusion Criteria:

General

* Insufficiently controlled diabetes mellitus in the judgment of the investigator
* Malignant tumor within the last 5 years with the exception of squamous and basal cell carcinoma or cervical carcinoma it situ
* Pregnancy, nursing, (or if fertile female) not willing to utilize birth control measures during study
* Unstable medical condition that is clinically significant in the judgment of the investigator: major organ system dysfunction

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 317 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of two doses of EVP-6124 (0.3, and 1.0 mg QD) versus placebo capsules (QD) for 84 days to subjects with schizophrenia who are on chronic stable atypical anti-psychotic therapy as determined by clinical safety and cognitive function. | 84 days

SECONDARY OUTCOMES:
Assessment of Clinical Efficacy | 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Chris Southard, Study Director — Syneos Health
Locations (29):
- United States (14):
  - Intergrated Medical and Behavioral Associates, Glendale, California
  - Excell Research, Oceanside, California
  - University of California, San Diego, San Diego, California
  - Affiliated Research Institute, San Diego, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Uptown Research Institute, Chicago, Illinois
  - Alexian Brothers Behavioral Health, Hoffman Estates, Illinois
  - CBH Health, LLC, Rockville, Maryland
  - CRI Worldwide, Willingboro, New Jersey
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - Vanderbilt Psychiatric Hospital, Nashville, Tennessee
  - FutureSearch Clinical Trials, L.P., Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
- Russia (5):
  - Arkhangelsk
  - Kazan'
  - Moscow
  - Saint Petersburg
  - Stavropol
- Serbia (5):
  - Clinical Site 1, Belgrade
  - Clinical Site 2, Belgrade
  - Clinical Site 3, Belgrade
  - Kragujevac
  - Niš
- Ukraine (5):
  - Crimea
  - Dnipro
  - Kiev
  - Odesa
  - Vinnytsia

REFERENCES:
- [Derived] Georgiades A, Davis VG, Atkins AS, Khan A, Walker TW, Loebel A, Haig G, Hilt DC, Dunayevich E, Umbricht D, Sand M, Keefe RSE. Psychometric characteristics of the MATRICS Consensus Cognitive Battery in a large pooled cohort of stable schizophrenia patients. Schizophr Res. 2017 Dec;190:172-179. doi: 10.1016/j.schres.2017.03.040. Epub 2017 Apr 20. PMID 28433500